CLINICAL TRIAL: NCT03432585
Title: Parent/Caregiver Conference Attendance Feasibility
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: American Society for Nutrition (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201800142
Record Dates: First submitted 2018-01-29; First posted 2018-02-14 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: feasibility; attendance; conference
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family Support Grant applicants: Participants include applicants for the Family Support Grants that will be provided for the American Society for Nutrition annual meeting who are willing to complete the applicant survey.
  Interventions: Behavioral: Applicant Survey

INTERVENTIONS:
Behavioral: Applicant Survey — This survey will ask a few brief demographic questions and will assess feedback from participants about preferences and barriers to conference attendance.

SUMMARY:
This study will assess and evaluate conference attendance feasibility and will gather feedback about preferences and barriers to attendance at the American Society for Nutrition annual conference.

DETAILED DESCRIPTION:
This study will use a survey provided on the American Society for Nutrition Family Support Grant application webpage for those who are registering to attend the American Society for Nutrition annual meeting and who are applying for this particular grant. The survey will take about 10 minutes to complete and will provide detailed information for assessment and evaluation of conference attendance feasibility and will also provide feedback about preferences and barriers related to attendance and this annual meeting.

ELIGIBILITY:
Inclusion Criteria:

* Must be an applicant for the Family Support Grant to the American Society for Nutrition annual conference that takes place in June 2018

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Applicants for the Family Support Grant to the American Society for Nutrition annual conference that takes place in June 2018
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Participant likelihood of attendance to the American Society for Nutrition annual meeting if provided with a family support grant | 20 minutes to complete survey
  5-point scale

SECONDARY OUTCOMES:
Grant option most likely to be used by participants | 20 minutes to complete survey
  4 options provided for participants to select. This will be tallied to determine which of the four options were most likely to be pursued.
Participants' opinion of greatest value of a family support grant should it be provided | 20 minutes to complete survey
  Participants will be asked to describe the greatest value of the family grant support. Potentially the top 7 selections will be recorded.
Participants' greatest barrier to attending the American Society for Nutrition annual meeting | 20 minutes to complete survey
  Participants will be asked to describe the greatest barrier to attending the American Society for Nutrition annual meeting. Potentially the top 10 selections will be recorded.
Most significant factor influencing the participant's decision to attend the American Society for Nutrition annual meeting | 20 minutes to complete survey
  Participants will be asked to describe the most significant factor influencing the participant's decision to attend the American Society for Nutrition annual meeting. Potentially the top 10 selections will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cardel, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cardel MI, Loop MS, Brown AW, Bohan Brown MM, Newsome F, Scott L, Lemas DJ, Krukowski RA. Implementation of a Family Support Grant to Subsidize Caregiving Needs and Support Attendance at American Society for Nutrition's Annual Professional Scientific Conference. Curr Dev Nutr. 2022 Jun 23;6(6):nzac076. doi: 10.1093/cdn/nzac076. eCollection 2022 Jun. PMID 35769451